CLINICAL TRIAL: NCT05329077
Title: A Study to Assess the Safety and Efficacy of Pulsenmore ES Home Ultrasound Device in Pregnant Women
Brief Title: Pulsenmore ES Device, Efficacy and Safety Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PulseNmore (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2201V1
Record Dates: First submitted 2022-03-20; First posted 2022-04-14 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-03

CONDITIONS: Perinatal Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Home Ultrasound users (Other): Single Arm home ultrasound in pregnant women users
  Interventions: Device: Pulsenmore ES home ultrasound device

INTERVENTIONS:
Device: Pulsenmore ES home ultrasound device — Pregnant participants will use Pulsenmore ES device to assess the safety and the efficacy of the device in monitoring fetal parameters

SUMMARY:
This is a multicenter, prospective, investigational device study designed to evaluate:

The safety, feasibility, and accuracy of the device, when used by pregnant individuals

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation.
* Gestational age >14 weeks with a prior scan demonstrating fetal viability and confirming dates.
* English or Spanish speaking.
* Ability to understand and sign the informed consent (available in English and Spanish).
* Ability to read and understand instructions that are required for equipment use (instructions available in both languages).

Exclusion Criteria:

* Multiple gestations.
* BMI >40.
* Known fetal and genetic anomalies.
* Subjects with skin problems in the abdominal area (such as wounds, cuts in the skin, and skin rash).
* Subjects allergic to the ultrasound probe materials.
* Non-English/ non-Spanish speaking.
* Unable to provide consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Comparison of device derived presence or absence of fetal cardiac activity to ground truth | Test to be conducted during week 14-38 of pregnancy
  The presence or absence of device derived fetal cardiac activity would be matched with the presence or absence of fetal cardiac activity derived by the ground truth (in-clinic ultrasound scan)
Comparison of device derived amniotic fluid level status, normal or abnormal, to ground truth | Test to be conducted during week 14-38 of pregnancy
  Comparison of device derived amniotic fluid level status, normal or abnormal, (measured by maximal vertical pocket in cm) would be matched with amniotic fluid level status derived from the ground truth (in-clinic ultrasound scan)

SECONDARY OUTCOMES:
Ability to assess fetal presentation from device derived input will be compared to the ground truth | Test to be conducted during week 14-38 of pregnancy
  Whether fetal presentation could be assessed or could not be assessed from device derived input compared to the input from ground truth (in-clinic ultrasound scan)
Ability to assess placental location from device derived input will be compared to the ground truth | Test to be conducted during week 14-38 of pregnancy
  Whether placental location could be assessed or could not be assessed from device derived input compared to the input from ground truth (in-clinic ultrasound scan)
Ability to detect fetal movement from device derived input will be compared to the ground truth | Test to be conducted during week 14-38 of pregnancy
  Whether fetal movement could be detected or could not be detected from device derived input compared to the input from ground truth (in-clinic ultrasound scan)
Ability to detect fetal breathing from device derived input will be compared to the ground truth | Test to be conducted during week >27-38 of pregnancy
  Whether fetal breathing could be detected or could not be detected from device derived input compared to the input from ground truth (in-clinic ultrasound scan)

CONTACTS AND LOCATIONS:
Overall Officials: Reem Abu-Rustum, MD, Principal Investigator — University of Florida
Locations (4):
- United States (4):
  - Center for Fetal Medicine and Women's Ultrasound, Los Angeles, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mount Sinai Hospital System, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guidelines for Perinatal Care, 8th Edition, AAP and ACOG 2017. ISBN: 978-1-934984-69-7 (ACOG)
- [Background] Abuhamad A, Zhao Y, Abuhamad S, Sinkovskaya E, Rao R, Kanaan C, Platt L. Standardized Six-Step Approach to the Performance of the Focused Basic Obstetric Ultrasound Examination. Am J Perinatol. 2016 Jan;33(1):90-8. doi: 10.1055/s-0035-1558828. Epub 2015 Aug 3. PMID 26238329